CLINICAL TRIAL: NCT02432729
Title: A Multi-center, Multi-region Smoking Cessation Study to Understand the Biological and Functional Changes Related to Smoking Cessation in Healthy Smokers Who Are Continuously Abstinent From Smoking for One Year
Brief Title: A Smoking Cessation Study to Understand the Biological and Functional Changes After One Year of Smoking Cessation
Acronym: RIBESC
Status: Completed | Type: Observational
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: SA-SCR-01; SA-SCR-01 (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2015-04-14; First posted 2015-05-04 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Cigarette Smoking
Keywords: smoking cessation; smoking abstinence; clinical, biological and functional changes; one year; healthy smokers; quit smoking
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine bio-banking samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Adult smokers who are willing to quit smoking within the next 30 days at the Screening Visit will be asked to continuously quit smoking for 1 year.
  Smokers who are not continuously abstinent from smoking or any nicotine/tobacco containing product from the actual quit date will be discontinued from the study.

SUMMARY:
The purpose of this study was to understand the biological and functional changes after one year of smoking cessation and to collect data on a broad range of biomarkers of exposure (BoExp) and biomarkers of effect (BoE).

DETAILED DESCRIPTION:
This was a 12 month, multi-region, multi-center, ambulatory study conducted in the US, Japan and Europe. Smokers who were willing to quit smoking within the next 30 days at the Screening Visit were enrolled to reach approximately 950 subjects continuously abstinent from smoking from Actual Quit Date (AQD) onwards at week 2, in order to achieve at least 190 successful quitters expected to complete the study. Once approximately 950 subjects reached week 2, screening and enrollment were stopped.

Compliance with smoking abstinence was verified by self-reporting, CO breath tests, and urine cotinine tests. Smokers who were not continuously abstinent from smoking [i.e., free from tobacco product use (e.g., CC, pipes, cigars, snus) or any nicotine-containing product (including electronic cigarettes) other than nicotine replacement therapy (NRT)] from their AQD onwards were discontinued from the study. At the end of the study, 358 subjects were verified as continuously abstinent from their AQD.

ELIGIBILITY:
Inclusion Criteria:

* Current healthy smoker as judged by the Principal Investigator(s) or designee(s).
* Subject is aged from 30 to 65 years old (inclusive).
* Subject has smoked for at least the last 10 years.
* Subject smoked more than 10 cigarettes/day on average over the last year.
* Subject is willing to quit smoking within the next 30 days.

Exclusion Criteria:

* Subject has clinically relevant medical conditions that in the opinion of the Investigators would jeopardize the safety of the participant or affect the validity of the study results.
* Subject has Forced Expiratory Volume in 1 second/Forced Vital Capacity(FEV1/FVC) < 0.7 and FEV1 < 80% predicted value at post-bronchodilator spirometry.
* Subject with FEV1/FVC < 0.75 (post-bronchodilator) and reversibility in FEV1 that is both > 12% and > 200 ml from pre- to post-bronchodilator values.
* Subject who took or is taking concomitant medication which may have an impact on the biomarkers of effect.
* Female subject is pregnant or is a breast-feeding.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, smoking subjects willing to quit smoking with no restriction on race and ethnicities will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Christel Contzen, MD, Principal Investigator — Synexus Clinical Research GmbH; Monika Tomaszewska-Kiecana, MD, Principal Investigator — BioVirtus Research Site Sp. z o.o.; Susannah Eyre, MD, Principal Investigator — Synexus, Merseyside Clinical Research Centre; Jed Rose, PhD, Principal Investigator — Rose Research Center; Koichi Nakamura, MD, Principal Investigator — Clinical Research Tokyo Hospital
Locations (5):
- Rose Research Center, Charlotte, North Carolina, United States
- Synexus Clinical Research GmbH, Frankfurt am Main, Hesse, Germany
- Clinical Research Tokyo Hospital, Tokyo, Japan
- BioVirtus Research Site Sp. z o.o., Kajetany, Poland
- Synexus, Merseyside Clinical Research Centre, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran CT, Felber Medlin L, Lama N, Taranu B, Ng W, Haziza C, Picavet P, Baker G, Ludicke F. Biological and Functional Changes in Healthy Adult Smokers Who Are Continuously Abstinent From Smoking for One Year: Protocol for a Prospective, Observational, Multicenter Cohort Study. JMIR Res Protoc. 2019 Jun 7;8(6):e12138. doi: 10.2196/12138. PMID 31199335
- [Result] Pouly, S., Haziza, C., Peck, M. J., & Peitsch, M. C. (2021). Clinical Assessment of ENDPs. In Toxicological Evaluation of Electronic Nicotine Delivery Products (pp. 385-459). Academic Press.

RESULTS

PARTICIPANT FLOW:
Groups:
- Abstinence3m Set: Enrolled subjects, who were abstinent from smoking from their actual quit date to at least Month 3, were included in the Abstinence3m set.
Period: Month 3 Visit
Arm/Group | Abstinence3m Set
Started | 720
Completed | 718
Not Completed | 2
Period: Month 6 Visit
Arm/Group | Abstinence3m Set
Started | 718
Completed | 632
Not Completed | 86
Period: Month 12 Visit
Arm/Group | Abstinence3m Set
Started | 632
Completed | 436
Not Completed | 196

BASELINE CHARACTERISTICS:
Population: All Regions
Groups:
- Enrolled: The Enrolled population included all subjects in the Full Safety Population, except 22 subjects enrolled at a site that was closed due to findings during a monitoring visit.
Arm/Group | Enrolled
Number analyzed (Participants) | 1184
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 591
  Male | 593
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 344
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 88
  White | 744
  More than one race | 3
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 73
  Ethnicity: Not Hispanic or Latino | 776
  Ethnicity: Japanese | 335
Weight [Mean (Standard Deviation); unit: kg] | 73.4 (14.9)
Height [Mean (Standard Deviation); unit: cm] | 170 (9.15)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (4.02)

OUTCOME MEASURES:

1. Primary Outcome: High Density Lipoprotein C (HDL-C).
Description: Concentrations of HDL-C measured in serum. Mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: Some subjects were prematurely discontinued from the study. Non-compliance with smoking abstinence was the most frequently reported reason for premature discontinuation from the study.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Abstinence3m: The Abstinence3m Set refers to enrolled subjects who were abstinent from smoking from their actual quit date to Month 3 (V8) or later.
Arm/Group | Abstinence3m
Number analyzed (Participants) | 720
mg/dL
  Baseline: number analyzed (Participants) | 710
  Baseline | 57.1 [55.8 to 58.4]
  Month 6: number analyzed (Participants) | 410
  Month 6 | 58.9 [57.1 to 60.7]
  Month 12: number analyzed (Participants) | 328
  Month 12 | 58.6 [56.6 to 60.5]

2. Primary Outcome: Low-density Lipoprotein Cholesterol (LDL-C)
Description: Concentrations of LDL-C measured in serum. Mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Abstinence3m Set: Enrolled subjects, who were abstinent from smoking from their actual quit date to Month 3, were included in the Abstinence3m set.
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
mg/dL
  Baseline: number analyzed (Participants) | 649
  Baseline | 131 [128 to 134]
  Month 6: number analyzed (Participants) | 440
  Month 6 | 136 [132 to 140]
  Month 12: number analyzed (Participants) | 355
  Month 12 | 138 [134 to 142]

3. Primary Outcome: Apo A1
Description: Concentrations of Apolipoprotein A1 measured in serum. Mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
mg/dL
  Baseline: number analyzed (Participants) | 710
  Baseline | 155 [153 to 158]
  Month 6: number analyzed (Participants) | 441
  Month 6 | 158 [155 to 161]
  Month 12: number analyzed (Participants) | 356
  Month 12 | 155 [152 to 158]

4. Primary Outcome: Apo B
Description: Concentrations of Apolipoprotein B measured in serum. Mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
mg/dL
  Baseline: number analyzed (Participants) | 712
  Baseline | 94.3 [92.4 to 96.2]
  Month 6: number analyzed (Participants) | 441
  Month 6 | 96.3 [93.8 to 98.7]
  Month 12: number analyzed (Participants) | 356
  Month 12 | 97.5 [94.8 to 100]

5. Primary Outcome: White Blood Cells (WBC).
Description: Concentrations of WBC measured in blood. Mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: GI/L
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
GI/L
  Baseline: number analyzed (Participants) | 717
  Baseline | 6.72 [6.58 to 6.86]
  Month 6: number analyzed (Participants) | 440
  Month 6 | 5.94 [5.79 to 6.09]
  Month 12: number analyzed (Participants) | 355
  Month 12 | 5.93 [5.75 to 6.11]

6. Primary Outcome: Hs-CRP
Description: Concentrations of high sensitivity C-reactive protein (hs-CRP) measured in serum. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
mg/L
  Baseline (mg/L): number analyzed (Participants) | 659
  Baseline (mg/L) | 0.856 [0.776 to 0.944]
  Month 6 (mg/L): number analyzed (Participants) | 441
  Month 6 (mg/L) | 0.841 [0.752 to 0.941]
  Month 12 (mg/L): number analyzed (Participants) | 356
  Month 12 (mg/L) | 0.963 [0.846 to 1.1]

7. Primary Outcome: Homocysteine
Description: Concentrations of Homocysteine measured in plasma. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
μmol/L
  Baseline (μmol/L): number analyzed (Participants) | 711
  Baseline (μmol/L) | 12.6 [12.3 to 12.9]
  Month 6 (μmol/L): number analyzed (Participants) | 442
  Month 6 (μmol/L) | 11.4 [11.1 to 11.8]
  Month 12 (μmol/L): number analyzed (Participants) | 356
  Month 12 (μmol/L) | 11.7 [11.3 to 12]

8. Primary Outcome: Fibrinogen
Description: Concentrations of Fibrinogen measured in plasma. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
mg/dL
  Baseline (mg/dL): number analyzed (Participants) | 645
  Baseline (mg/dL) | 326 [321 to 331]
  Month 6 (mg/dL): number analyzed (Participants) | 424
  Month 6 (mg/dL) | 310 [304 to 316]
  Month 12 (mg/dL): number analyzed (Participants) | 348
  Month 12 (mg/dL) | 312 [305 to 319]

9. Primary Outcome: Platelets
Description: Concentrations of Platelets measured in plasma. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: GI/L
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
GI/L
  Baseline (GI/L): number analyzed (Participants) | 717
  Baseline (GI/L) | 239 [235 to 243]
  Month 6 (GI/L): number analyzed (Participants) | 439
  Month 6 (GI/L) | 240 [235 to 245]
  Month 12 (GI/L): number analyzed (Participants) | 352
  Month 12 (GI/L) | 241 [236 to 246]

10. Primary Outcome: 11-dehydrothromboxane B2 (11-DTXB2).
Description: Concentrations measured in urine and expressed as concentration adjusted for creatinine. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
pg/mg creat
  Baseline (pg/mg creat): number analyzed (Participants) | 543
  Baseline (pg/mg creat) | 572 [546 to 601]
  Month 6 (pg/mg creat): number analyzed (Participants) | 437
  Month 6 (pg/mg creat) | 433 [409 to 458]
  Month 12 (pg/mg creat): number analyzed (Participants) | 352
  Month 12 (pg/mg creat) | 436 [411 to 463]

11. Primary Outcome: 8-epi-prostaglandin F2α (8-epi-PGF2α).
Description: Concentrations of 8-epi-PGF2α measured in urine and expressed as concentration adjusted for creatinine. Geometric Means are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
pg/mg creat
  Baseline (pg/mg creat): number analyzed (Participants) | 548
  Baseline (pg/mg creat) | 242 [233 to 251]
  Month 6 (pg/mg creat): number analyzed (Participants) | 443
  Month 6 (pg/mg creat) | 199 [190 to 207]
  Month 12 (pg/mg creat): number analyzed (Participants) | 357
  Month 12 (pg/mg creat) | 189 [180 to 197]

12. Primary Outcome: MPO
Description: Concentrations of Myeloperoxidase measured in serum. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/L
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
μg/L
  Baseline (μg/L): number analyzed (Participants) | 716
  Baseline (μg/L) | 133 [126 to 140]
  Month 6 (μg/L): number analyzed (Participants) | 442
  Month 6 (μg/L) | 144 [133 to 155]
  Month 12 (μg/L): number analyzed (Participants) | 356
  Month 12 (μg/L) | 202 [187 to 217]

13. Primary Outcome: Soluble Intercellular Adhesion Molecule 1 (sICAM-1).
Description: Concentrations of sICAM-1 measured in serum. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
ng/mL
  Baseline (ng/mL): number analyzed (Participants) | 661
  Baseline (ng/mL) | 229 [223 to 236]
  Month 6 (ng/mL): number analyzed (Participants) | 442
  Month 6 (ng/mL) | 201 [195 to 207]
  Month 12 (ng/mL): number analyzed (Participants) | 356
  Month 12 (ng/mL) | 194 [187 to 200]

14. Primary Outcome: Albumin
Description: Concentrations of Albumin measured in urine and expressed as concentration adjusted for creatinine. Geometric mean values are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g creat
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
mg/g creat
  Baseline (mg/g creat): number analyzed (Participants) | 579
  Baseline (mg/g creat) | 5.68 [5.36 to 6.03]
  Month 6 (mg/g creat): number analyzed (Participants) | 443
  Month 6 (mg/g creat) | 5.69 [5.28 to 6.13]
  Month 12 (mg/g creat): number analyzed (Participants) | 356
  Month 12 (mg/g creat) | 5.51 [5.12 to 5.94]

15. Primary Outcome: Carboxyhemoglobin (COHb).
Description: Carboxyhemoglobin (COHb) is assayed from whole blood. Expressed as % of saturation of hemoglobin. Geometric means are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percentage
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
percentage
  Baseline: number analyzed (Participants) | 424
  Baseline | 2.78 [2.61 to 2.96]
  Month 6: number analyzed (Participants) | 417
  Month 6 | 0.724 [0.664 to 0.789]
  Month 12: number analyzed (Participants) | 352
  Month 12 | 0.758 [0.691 to 0.831]

16. Primary Outcome: HbA1c
Description: Glycosylated hemoglobin (HbA1c) is assayed from whole blood. Geometric means are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
percentage of glycated hemoglobin
  Baseline: number analyzed (Participants) | 713
  Baseline | 5.42 [5.39 to 5.44]
  Month 6: number analyzed (Participants) | 439
  Month 6 | 5.39 [5.36 to 5.42]
  Month 12: number analyzed (Participants) | 354
  Month 12 | 5.45 [5.42 to 5.49]

17. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1), Pre-bronchodilator and Expressed as Percentage Predicted (FEV1 %Pred).
Description: FEV1 pre-bronchodilator and expressed as percentage predicted (FEV1 %pred).
  Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced expiratory volume (FEV) in one second is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FEV1
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
Percent of predicted FEV1
  Baseline: number analyzed (Participants) | 674
  Baseline | 94.5 [93.7 to 95.4]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 94.2 [93.1 to 95.4]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 93.9 [92.6 to 95.3]

18. Primary Outcome: FEV1 Post-bronchodilator and Expressed as Percentage Predicted (FEV1 %Pred).
Description: FEV1 post-bronchodilator and expressed as percentage predicted (FEV1 %pred). Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced expiratory volume (FEV) in one second is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FEV1
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
Percent of predicted FEV1
  Baseline: number analyzed (Participants) | 673
  Baseline | 97.1 [96.2 to 98]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 96.7 [95.6 to 97.9]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 96.5 [95.2 to 97.8]

19. Primary Outcome: Forced Vital Capacity (FVC) Pre-bronchodilator, Expressed as Percentage Predicted (FVC %Pred).
Description: Pre-bronchodilator Forced Vital Capacity, expressed as percentage predicted (FVC %pred). Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced vital capacity (FVC) is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FVC
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
Percent of predicted FVC
  Baseline: number analyzed (Participants) | 674
  Baseline | 101 [99.7 to 101]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 100 [99 to 101]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 99.1 [97.8 to 100]

20. Primary Outcome: FVC Post-bronchodilator, Expressed as Percentage Predicted (FVC %Pred).
Description: Post-bronchodilator Forced Vital Capacity, expressed as percentage predicted (FVC %pred). Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced vital capacity (FVC) is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FVC
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
Percent of predicted FVC
  Baseline: number analyzed (Participants) | 673
  Baseline | 100 [99.1 to 101]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 99.5 [98.3 to 101]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 98.6 [97.3 to 99.9]

21. Primary Outcome: FEV1/FVC Pre-bronchodilator Expressed as a Ratio
Description: Pre-bronchodilator FEV1/FVC expressed as a ratio. Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced vital capacity (FVC) is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration, and the forced expiratory volume (FEV) in one second is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
ratio
  Baseline: number analyzed (Participants) | 674
  Baseline | 0.771 [0.766 to 0.776]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 0.77 [0.764 to 0.776]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 0.778 [0.772 to 0.785]

22. Primary Outcome: FEV1/FVC Post-bronchodilator Expressed as a Ratio
Description: Post-bronchodilator FEV1/FVC expressed as a ratio. Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The primary signal measured in spirometry may be volume or flow. The forced vital capacity (FVC) is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration, and the forced expiratory volume (FEV) in one second is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
ratio
  Baseline: number analyzed (Participants) | 673
  Baseline | 0.796 [0.791 to 0.8]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 0.797 [0.791 to 0.802]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 0.803 [0.797 to 0.809]

23. Primary Outcome: FEF 25-75 Forced Expiratory Flow, Pre-bronchodilator, Expressed as Percentage Predicted (FEF 25-75 %Pred)
Description: Pre-bronchodilator FEF 25-75, expressed as percentage predicted (FEF 25-75 %pred). Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The forced expiratory flow between 25% and 75% of the FVC (FEF25-75%) is defined as the forced expiratory flow during the middle half of the FVC; the average flow from the point at which 25% of the FVC has been exhaled to the point at which 75% of the FVC has been exhaled.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FEF 25-75%
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
Percent of predicted FEF 25-75%
  Baseline: number analyzed (Participants) | 674
  Baseline | 84.8 [82.9 to 86.7]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 84.2 [81.8 to 86.6]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 86.6 [84 to 89.3]

24. Primary Outcome: FEF 25-75 Forced Expiratory Flow, Post-bronchodilator, Expressed as Percentage Predicted (FEF 25-75 %Pred)
Description: Post-bronchodilator FEF 25-75, expressed as percentage predicted (FEF 25-75 %pred). Mean values are provided as descriptive statistics.
  Spirometry is a physiological test that measures how an individual inhales or exhales volumes of air as a function of time. The forced expiratory flow between 25% and 75% of the FVC (FEF25-75%) is defined as the forced expiratory flow during the middle half of the FVC; the average flow from the point at which 25% of the FVC has been exhaled to the point at which 75% of the FVC has been exhaled.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FEF 25-75%
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
Percent of predicted FEF 25-75%
  Baseline: number analyzed (Participants) | 673
  Baseline | 95.7 [93.7 to 97.7]
  Month 6: number analyzed (Participants) | 437
  Month 6 | 95.8 [93.9 to 98.3]
  Month 12: number analyzed (Participants) | 334
  Month 12 | 98.1 [95.4 to 101]

25. Primary Outcome: Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL).
Description: Concentrations of Total NNAL measured in urine and expressed as concentration adjusted for creatinine. Geometric means are provided as descriptive statistics.
Time Frame: Baseline; 6 month; 12 month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | Abstinence3m Set
Number analyzed (Participants) | 720
pg/mg creat
  Baseline (pg/mg creat): number analyzed (Participants) | 585
  Baseline (pg/mg creat) | 125 [114 to 136]
  Month 6 (pg/mg creat): number analyzed (Participants) | 443
  Month 6 (pg/mg creat) | 5.11 [4.68 to 5.58]
  Month 12 (pg/mg creat): number analyzed (Participants) | 357
  Month 12 (pg/mg creat) | 4.37 [3.99 to 4.78]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, for a duration of up to 66 weeks for each subject.
Groups:
- Enrolled Population: The Enrolled Population included 1184 subjects enrolled from the screened population.
Arm/Group | Enrolled Population
All-Cause Mortality (participants affected / at risk) | 1/1184
Serious Adverse Events (participants affected / at risk) | 17/1184
Other Adverse Events (participants affected / at risk) | 313/1184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Population (N=1184)
Pyelonephritis (Infections and infestations) | 2 (5)
Pneumonia (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (4)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Population (N=1184)
Nasopharyngitis (Infections and infestations) | 158 (213)
Upper respiratory tract infection (Infections and infestations) | 83 (94)
Weight increased (Investigations) | 72 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT02432729/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02432729/SAP_001.pdf